CLINICAL TRIAL: NCT02848586
Title: Effects of E-cigarettes (ECIGs) on Pulmonary Inflammation and Behavior in HIV Infected Smokers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment failed due to lack of subjects meeting the eligibility criteria
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00066481; P30AI064518 (NIH)
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2019-12

CONDITIONS: Lung Inflammation; HIV Seropositivity
Keywords: HIV; ECIGS; e-cigarettes; lung inflammation
MeSH Terms: conditions — Pneumonia; HIV Seropositivity; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECIGS (Active Comparator): Subjects will receive e-cigarettes for a total of 4 weeks. A mobile contingency management (mCM) procedure will be used to provide monetary reinforcement for biochemically verified abstinence from combustible cigarettes. After 4 weeks, subjects will be allowed to transition back to their chosen combustible cigarette product for an additional 2 weeks. Respiratory assessments will occur at study arm assignment (Visit 1) to establish baseline measures of lung function, oxidative stress, and systemic inflammation, repeated again 4 weeks after transition to ECIG (Visit 4) and again 2 weeks after stopping ECIG (Visit 5). Neuro-cognitive and behavioral assessments will occur at Visits 2, 3, 4 and 5.
  Interventions: Other: ECIGS; Behavioral: mobile contingency management (mCM)
- Usual brand (Active Comparator): Subjects will receive their usual brand of combustible cigarettes for a total of 4 weeks. A mobile contingency management mCM procedure will be used. Respiratory assessments will occur at study arm assignment (Visit 1) to establish baseline measures of lung function, oxidative stress, and systemic inflammation, repeated again 4 weeks later (Visit 4) and again 2 weeks later (Visit 5). Neuro-cognitive and behavioral assessments will occur at Visits 2, 3, 4 and 5.
  Interventions: Behavioral: mobile contingency management (mCM); Other: Usual brand

INTERVENTIONS:
Other: ECIGS — 15 subjects will receive ECIGs and 5 control subjects will continue to smoke their chosen usual brand of combustible cigarettes (UB). Each group will receive either ECIG or UB for a total of 4 weeks and undergo pulmonary and behavioral assessments during this period. A mobile contingency management (mCM) procedure will be used to provide monetary reinforcement for biochemically verified abstinence from combustible cigarettes. Participants in the UB group will also undergo mCM procedures, but contingencies will differ. After 4 weeks, the ECIG group will be allowed to transition back to their chosen combustible cigarette product for an additional 2 weeks with additional pulmonary and behavioral assessments. All subjects will undergo three respiratory assessments in the DCRU.
  Other Names: Port Royale
  Arms: ECIGS
Behavioral: mobile contingency management (mCM) — mCM procedures are a novel smoking cessation tool previously used in the field by our colleagues in the Beckham research group. This equipment is part of a procedure called "mobile contingency management" or "mCM". The participant will use a study smartphone to record his/her CO levels and moods at random times of the day and to verify his/her cigarette usage. The mCM program will reward the participant for each CO level and data transmitted to the study team. The study team will provide detailed information and training to allow them to participate in this part of the study.
Other: Usual brand — The usual brand of cigarettes is the control group in this study. 5 participants will be allowed to continue using their "usual brand" of combustible cigarette in this arm of the study.
  Arms: Usual brand

SUMMARY:
The purpose of this study is to determine if using e-cigarettes (ECIG) rather than regular tobacco cigarettes alters lung inflammation in people with and without HIV. The study is also interested in asking subjects their opinion on the use of ECIG and how they make them feel. This study is for research purposes only and is not intended to treat asthma or HIV or to modify tobacco use.

DETAILED DESCRIPTION:
Title: Effects of e-cigarettes (ECIGs) on pulmonary inflammation and behavior in HIV infected smokers

Purpose of the Study: Even though smoking is the leading cause of preventable disease and deaths in the U.S., millions of Americans continue to smoke cigarettes, including 16% of persons in the general population and 40-70% of all HIV-infected patients. In contrast to the relatively known adverse effects of combustible cigarettes, the rapid emergence of e-cigarettes have raised numerous questions regarding their health effects which may be amplified in vulnerable populations and those already immunocompromised such as HIV-infected patients. The goal of the proposed research is to gain an understanding of the cellular and inflammatory mechanisms that occur in the lung of HIV-infected smokers who transition from conventional tobacco cigarettes to e-cigarettes and to characterize their behavioral and neurocognitive effects. These efforts will provide first in kind data on the effects of ECIGs in this study population and provide valuable data to develop needed regulatory policies.

Background & Significance: While rates of cigarette smoking are gradually decreasing in the US, the burden of tobacco abuse among people living with HIV remains undisputedly high with prevalence estimates two to three times higher than the general population (42.4% vs. 16%). Although ECIGs likely contain significantly fewer numbers of toxicants compared to combustible cigarettes, it is not yet clear whether ECIG are less harmful than their traditional tobacco counterparts and what, if any, effects they have on behavior and neurocognitive functioning. The biological effects of ECIG on lung health have not yet been sufficiently characterized due the relatively nascent nature of the field. While combustible tobacco use induces oxidant stress in the airways of healthy smokers, little work to date has established the effect of ECIG use on oxidant stress in human airways. Transitioning the smoker from combustible tobacco to ECIG may decrease lung oxidative stress, improve lung function and decrease withdrawal symptoms and deficits in neurocognition commonly seen with tobacco withdrawal.

Design & Procedures: 15 HIV-infected adults will be recruited from the Duke Infectious Diseases Clinic. In addition, 5 HIV-negative adults will be recruited from the community through flyers. For this pilot study, 15 willing subjects will receive ECIGs and 5 control subjects will continue to smoke their chosen usual brand of combustible cigarettes (UB). Each group will receive either ECIG or UB for a total of 4 weeks and undergo pulmonary and behavioral assessments during this period. In order to examine pulmonary and behavioral effects of ECIG in the absence of combustible cigarette use, a mobile contingency management (mCM) procedure will be used to provide monetary reinforcement for biochemically verified discontinuation of the use of combustible cigarettes. Participants in the UB group will also undergo mCM procedures, but contingencies will differ. After 4 weeks, the ECIG group will be allowed to transition back to their chosen combustible cigarette product for an additional 2 weeks with additional pulmonary and behavioral assessments. All subjects will undergo three respiratory assessments in the Duke Clinical Research Unit (DCRU). The first respiratory assessment will occur at study arm assignment (V1) to establish baseline measures of lung function, oxidative stress, and systemic inflammation. Pulmonary assessments will be repeated again 4 weeks after transition to ECIG or continued UB use (V4). A final respiratory assessment (V5) will occur 2 weeks after stopping ECIG or after 6 weeks of continued UB use to measure changes relative to baseline lung function, oxidative stress, and inflammation. Neuro-cognitive and behavioral visits will take place in Duke South or at the Center for Addiction Science and Technology (CfAST) and occur at Visit 2 (mCM transition), and respiratory visits (V4 & V5) as well as 2 weeks after ECIG transition/ continued UB use (V3)

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported smoking of ≥10 cigarettes/day for >2yrs
2. Smoke regular filtered cigarettes or machine-rolled cigarettes with a filter
3. Have expired CO concentrations of ≥10ppm or morning urinary cotinine >100ng/ml (as measured with NicAlert)

   * If present in the afternoon with CO concentration >10ppm then no cotinine test
   * If less than <10 then urinary continine
4. No serious quit attempt in the prior 3 months. This includes use of any FDA approved smoking cessation medication (varenicline, bupropion [used specifically as a quitting aid], patch, gum, lozenge, inhaler, and nasal spray) in the past 3 months as an indication of treatment seeking
5. No plans to quit in the next 3 months (set quit date, designated method, etc.)
6. Participants must be interested in substituting their normal combustible tobacco products with ECIG for 4 weeks
7. Willing and able to give informed consent and adhere to visit/protocol schedules
8. Reported method of birth control for at least 3 months prior to enrollment for women of child bearing potential
9. Read and write in English

   HIV-positive patients must meet the following additional inclusion criteria:
10. Currently receive HIV care at the Duke Infectious Diseases Clinic
11. Receiving stable ART treatment (i.e., no ART class changes or changes in dose in response to poor virological control) for >9 months with viral loads <200 copies/mL

Exclusion Criteria:

1. Alcohol intoxication measured by positive BAL (any detectable level)
2. Acute psychiatric symptoms (e.g. mania, hallucinations) preventing completion of the study procedures
3. Current use of nicotine replacement or other pharmacotherapy for smoking cessation
4. Positive pregnancy test for women (pregnant women will be referred for smoking cessation) and/or nursing women
5. Use of other tobacco products (e.g. chew tobacco, snuff) on >10 of the past 30 days will exclude patients to ensure they are primarily cigarette smokers
6. Use of hand-rolled, roll your own cigarettes
7. Use of marijuana or cigars >2 times/week will be excluded from the study. Subjects using marijuana ≤2 times/week will be required to refrain for the duration of the protocol.
8. Positive urine drug screen other than marijuana or currently prescribed medications.
9. Known allergy to propylene glycol or vegetable glycerin (potential constituents of ECIG)
10. Use of an ECIG for 5 or more within 30 days or any use in the past 7 days
11. Patients with a formal clinical or spirometry diagnosis of co-existing inflammatory airway conditions of COPD and/or asthma or underlying illnesses that may result in altered lung function (bronchiectasis, prior surgical lung resection, extensive cavitary infectious disease, etc.)
12. An ED visit or inpatient admission for a primary respiratory diagnosis or treatment with antibiotics within 60 days of enrollment
13. History of any systemic or inhaled corticosteroids within 3 months
14. Regular substance abuse or inpatient treatment for these in the past 6 months
15. Poorly controlled concomitant conditions that pose additional procedure risk as determined by the investigator

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Changes in sputum glutathione concentration | Weeks 1, 6, and 8
  Sputum will be obtained by each participant and a sputum supernatant prepared. Glutathione concentration will be measured in the sputum supernatant.

SECONDARY OUTCOMES:
Change in sputum 8-isoprostane | Weeks 1, 6, and 8
Change in nitrate/nitrite | Weeks 1, 6, and 8
Change in sputum inflammatory cytokines | Weeks 1, 6, and 8
Change in withdrawal, as measured by questionnaire | Weeks 1, 2, 4, 6, 8
Change in craving, as measured by questionnaire | Weeks 1, 2, 4, 6, 8
Change in neurocognition, as measured by questionnaire | Weeks 2, 6, 8

CONTACTS AND LOCATIONS:
Overall Officials: David Murdoch, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No